CLINICAL TRIAL: NCT01282099
Title: Is There a Canary in the PICU? A Critical Appraisal of the Role of Near Infrared Spectroscopy (NIRS) in the Pediatric Intensive Care Unit (PICU)
Brief Title: A Critical Appraisal of the Role of Near Infrared Spectroscopy (NIRS) in the Pediatric Intensive Care Unit (PICU)
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 100603
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Pediatric Intensive Care Unit
Keywords: all children entering the PICU eligible for enrollment; age range: neonate to 16 years

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiac patients: Postoperative congenital heart disease patients requiring stay in the PICU
- non-cardiac patients: non-cardiac patients requiring stay in the PICU

SUMMARY:
While near infrared spectroscopy is an exciting technology, scientific rigor is required in order to optimize its appropriate use in the clinical arena. This study will explore the feasibility and clinical applicability of data obtained from the NIRS device. The ability to noninvasively monitor peripheral perfusion remains an area of intense research. The most widely used method is pulse oximetry. The international mandate of its use in operating rooms in the early 1990s after the publication of the Harvard minimum standards for monitoring speaks to its unquestionable utility. Its pervasive application notwithstanding, pulse oximetry merely provides a calibrated ratio of arterial and venous hemoglobin saturation. While this data is valuable, time-tested, and even may hold the promise of accurately noninvasively trending cardiac output, cellular dysmetabolism -- hallmarks of vulnerable, yet viable tissue beds -- are beyond the predictive values of currently available devices.

ELIGIBILITY:
Inclusion Criteria:

* neonates to 16 year olds
* requiring stay in the PICU greater than 24 hours

Exclusion Criteria:

* anticipated PICU stay less than 24 hours
* children with ALLOW NATURAL DEATH orders

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: neonates to 16 years of age requiring stay in the PICU postoperative congenital heart disease patients non-cardiac patients
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Comparison of data obtained using Near Infrared Spectroscopy (NIRS) versus traditional Pediatric Intensive Care Unit (PICU) clinical parameters | 48 hours
  Upon arrival to PICU, 1 lead will be place on the forehead to monitor cerebral regional saturation (CrSO2)and 1 lead will be placed on the flank to measure somatic regional saturation (SrSO2).

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Forbes, MD, FAAP, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Lima A, Bakker J. Noninvasive monitoring of peripheral perfusion. Intensive Care Med. 2005 Oct;31(10):1316-26. doi: 10.1007/s00134-005-2790-2. Epub 2005 Sep 17. PMID 16170543
- [Background] Kelleher JF. Pulse oximetry. J Clin Monit. 1989 Jan;5(1):37-62. doi: 10.1007/BF01618369. PMID 2647912
- [Background] Webster JG 1997 Design of Pulse Oximeters (Bristol: Institute of Physics Publishing)
- [Background] Lima AP, Beelen P, Bakker J. Use of a peripheral perfusion index derived from the pulse oximetry signal as a noninvasive indicator of perfusion. Crit Care Med. 2002 Jun;30(6):1210-3. doi: 10.1097/00003246-200206000-00006. PMID 12072670
- [Background] Armonda RA, McGee B, Veznadaraglu E, Rosenwasser RH. Near-infrared spectroscopy (NIRS) measurements of cerebral oximetry in the neurovascular ICU. Crit Care Med 1999; 27:173
- [Background] Kohn, Linda T, Corrigan, J, Donaldson, Molla S. To err is human: building a safer health system. Institute of Medicine (U.S.). Committee on Quality of Health Care in America. Vol. 627, Nov.1999
- [Background] Standards of evidence for the safety and effectiveness of critical care monitoring devices and related interventions. Coalition for Critical Care Excellence: Consensus Conference on Physiologic Monitoring Devices. Crit Care Med. 1995 Oct;23(10):1756-63. doi: 10.1097/00003246-199510000-00022. PMID 7587243
- [Background] Prough DS, Pollard V. Cerebral near-infrared spectroscopy: ready for prime time? Crit Care Med. 1995 Oct;23(10):1624-6. doi: 10.1097/00003246-199510000-00004. No abstract available. PMID 7587225
- [Background] Feldman MD, Petersen AJ, Karliner LS, Tice JA. Who is responsible for evaluating the safety and effectiveness of medical devices? The role of independent technology assessment. J Gen Intern Med. 2008 Jan;23 Suppl 1(Suppl 1):57-63. doi: 10.1007/s11606-007-0275-4. PMID 18095046
- [Background] Mullner M, Sterz F, Binder M, Hirschl MM, Janata K, Laggner AN. Near infrared spectroscopy during and after cardiac arrest--preliminary results. Clin Intensive Care. 1995;6(3):107-11. PMID 10150558
- [Background] Schwarz G, Litscher G, Kleinert R, Jobstmann R. Cerebral oximetry in dead subjects. J Neurosurg Anesthesiol. 1996 Jul;8(3):189-93. doi: 10.1097/00008506-199607000-00001. PMID 8803829
- [Background] Tobias JD. Cerebral oximetry monitoring with near infrared spectroscopy detects alterations in oxygenation before pulse oximetry. J Intensive Care Med. 2008 Nov-Dec;23(6):384-8. doi: 10.1177/0885066608324380. PMID 18794168
- [Background] Tobias JD. Cerebral oximetry monitoring provides early warning of hypercyanotic spells in an infant with tetralogy of Fallot. J Intensive Care Med. 2007 Mar-Apr;22(2):118-20. doi: 10.1177/0885066606297966. PMID 17456731
- [Background] Lee TS, Hines GL, Feuerman M. Significant correlation between cerebral oximetry and carotid stump pressure during carotid endarterectomy. Ann Vasc Surg. 2008 Jan;22(1):58-62. doi: 10.1016/j.avsg.2007.07.022. Epub 2007 Nov 26. PMID 18023554